CLINICAL TRIAL: NCT04510116
Title: Preventing Alcohol Use Among African American Youths
Brief Title: Adults In The Making Prevention Trial
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Gene H. Brody, Regents Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-10106
Record Dates: First submitted 2020-08-04; First posted 2020-08-12 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIM preventive intervention (Experimental): Families were assigned to receive a 6 session, 12 hour prevention program in their community.
  Interventions: Behavioral: Adults in the Making program
- Control (No Intervention): Families were assigned to no intervention control.

INTERVENTIONS:
Behavioral: Adults in the Making program — The AIM prevention program, modeled after an existing family-based skills-training intervention in a group format for rural African American preadolescents, consists of six consecutive weekly group meetings held at community facilities, with separate parent and youth skill-building curricula and a family curriculum. Each of the six meetings includes separate, concurrent training sessions for parents and youth, followed by a joint parent-youth session during which the families practice the skills they learned in their separate sessions. Concurrent and family sessions each last 1 hour. Thus, both parents and youth receive 12 hours of prevention training.
  Other Names: AIM
  Arms: AIM preventive intervention

SUMMARY:
This study was a randomized prevention trial investigating the efficacy of the Adults in the Making (AIM) prevention program against a control condition. The primary outcome variable is alcohol use. The study sample were 367 African American seniors in high school and their primary caregivers. The AIM program is a 6 session (12 hour) family-centered intervention designed to deter alcohol use.

DETAILED DESCRIPTION:
The study investigators designed a multicomponent prevention program to deter substance use among African American emerging adults in rural Georgia (SAAF-Emerging Adult Program, SAAF-EAP). The intervention's delivery is modeled after an existing prevention program designed by Dr. Brody called, The Strong African American Families (SAAF) program and included a series of separate weekly sessions for emerging adults, their parents, and extended family members, as well as sessions in which participants interact with one another to apply the skills learned in the separate sessions. The sample consisted of 690 families with a high school senior, half of whom will be assigned randomly to a prevention group and half of whom will be assigned to a control group. Pre-intervention, post-intervention, and follow-up assessments of emerging adults' substance use were conducted with the entire sample. The study started when the participants were high school seniors, and followed them and their families as the youths enter emerging adulthood. The conceptual model that guided the program incorporated the following predictors: (1) autonomy-promoting parenting and responsive family relationships, characterized by developmentally appropriate instrumental and emotional support, expectations and discussions about emerging adults' roles and responsibilities, affectively positive relationships that feature open communication, and adaptive racial socialization that includes strategies for dealing with discrimination; (2) contextual stressors, including racial discrimination, poverty, and limitations in educational and occupational opportunities; (3) negative emotions and the avoidant coping responses they elicit; (4) emerging adults' future orientation, self-regulation, emotion regulation, racial identity, and sense of adult status; (5) affiliations with substance-using friends and romantic partners; and (6) cognitive antecedents of substance use, including prototypes of substance-using agemates and willingness to use substances in risk-conducive situations. To examine these constructs, the investigators implemented a multi-informant design that included assessments from emerging adults, their friends and romantic partners, their primary caregivers, and their extended family members.

ELIGIBILITY:
Inclusion Criteria:

* Residence in county where sampling was targeted
* Youth self identified as African American or Black

Exclusion Criteria:

* Unable to complete survey measures or participate in intervention due to mental health concerns

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 367 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Alcohol use | follow up at 27 months post baseline
  Past month frequency of alcohol use, item from Monitoring the Future Survey
Conduct problems | follow up at 27 months post baseline
  Parent reported rule breaking and aggression sub-scales of the Child Behavior Checklist. The combined subscales yield a score ranging from 0-38 with higher scores indicating more conduct problems

SECONDARY OUTCOMES:
Depressive symptoms | follow up at 27 months post baseline
  parent reported depressed/anxious symptoms on a subscale of the Child Behavor Checklist that ranged from 0-24 with higher scores indicating more depressive or anxiety symptoms
Protective caregiving | follow up at 6 months post baseline
  parent reported scale assessed the extent to which the primary caregiver provided emotional support, was accessible to the youth, and discussed difficult issues with which the youth was dealing. The 15 item scale ranged from 15-60 with higher scores reflecting more protective caregiving.

CONTACTS AND LOCATIONS:
Overall Officials: Gene Brody, PhD, Principal Investigator — University of Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brody GH, Yu T, Chen E, Miller GE, Barton AW, Kogan SM. Family-Centered Prevention Effects on the Association Between Racial Discrimination and Mental Health in Black Adolescents: Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 Mar 1;4(3):e211964. doi: 10.1001/jamanetworkopen.2021.1964. PMID 33760092